CLINICAL TRIAL: NCT02248909
Title: Non-interventional Multicenter Study of Spirometry Use to Diagnose COPD and to Prescribe Treatment to COPD Patients in the Outpatient Institutions of the healthcaRe System of the Russian FederaTion
Brief Title: Non-interventional Study of Spirometry Use to Diagnose COPD (Chronic Obstructive Pulmonary Disease) and to Prescribe Treatment to COPD Patients in the Outpatient Institutions
Acronym: SUPPORT
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RRU-XXX-2014/2
Record Dates: First submitted 2014-09-19; First posted 2014-09-25 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-01

CONDITIONS: COPD
Keywords: COPD, Primary Care, Spirometry, Risk factors
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with COPD risk factors: Group of subjects with COPD risk factors. This group will include patients aged ≥40 years, with smoking history of ≥10 pack years and long-active (not less than 3 consequent months) respiratory complaints
- Patients previously diagnosed with COPD: Group of patients who according to the medical records have already been diagnosed with COPD

SUMMARY:
This study is an observational multicenter descriptive study. The study will be conducted in primary outpatient medical institutions in different cities of the RF. Primary care doctors who are primary contact for greater part of the population in RF including COPD patients will be invited as investigators. This observational descriptive study will be conducted within the routine practice of outpatient institutions. Since spirometry is not an integral part of the current all-round clinical practice, only those sites where spirometry test is routinely used in examination of patients with COPD risk factors and when monitoring condition of COPD patients will take part in the study. Thus the decision about spirometry in every study subject will be determined only by the existing treatment approaches.

DETAILED DESCRIPTION:
The study is an observational multicenter descriptive study. No hypothesis is checked in the study.

3000 patients with COPD risk factors are planned to be enrolled into the study (current smokers and former smokers with smoking history of ≥10 pack/years at the age of >40 years who have respiratory complaints) and 1450 patients previously diagnosed with COPD who contacted the physicians of outpatient institutions during the study (for 3 months) and are currently in remission.

100 patients with COPD risk factors and approximately 50 patients early diagnosed with COPD currently being stable are planned to be enrolled in each site.

Physicians and pulmonologists of the outpatient institutions of the Russian Federation will take part in the study in about 30 sites in 18 cities (a total of 31% of RF population live in the cities).

The observational descriptive study will be conducted within the routine practice of outpatient institutions. Examining and treatment of patients will be performed according to the rules of the routine practice.

Patients will be enrolled into the study as they visit the outpatient institutions for the medical care. The study does not imply any special invitation of COPD patients to the sites for them to be enrolled into the study. Therefore the conditions are made for the study population to reflect the typical visitors of the primary care medical institutions in different RF (Russian Federation) regions. Patients are enrolled into the study regardless the reason for appointment with a doctor. A reason for the appointment can be respiratory complaints as well as any other diseases or certificates and conclusions. To be enrolled into the study the subjects must sign the written Informed Consent Form (ICF) to participate in the study and to use personal data confidentially.

To investigate the role of spirometry in diagnostics and management of the COPD patients, two groups of patients are supposed to be included into the study.

ELIGIBILITY:
Patients with COPD risk factors must meet all the following inclusion criteria:

1. Age ≥ 40 years.
2. Smoker or former smoker with smoking history of ≥ 10 pack years (patient is considered to be a former smoker in case of smoking cessation for ≥6 months) (the patient smokes or smoked before but then gave up smoking. The obligatory condition: smoking history is ≥10 pack years. It means that the patient smoked a pack per day for 10 years or half a pack for 20 years or 2 packs a day for 5 years).
3. Any complaints judged by the investigator to be possibly related to the respiratory diseases (chronic cough, dyspnea, cough with sputum, feeling of stiffness in the chest) or the evidence of the chronic respiratory diseases (chronic bronchitis in remission, pneumosclerosis) in the medical chart.
4. The patient is expected to have the spirometry test performed in accordance with the current medical practice before inviting him to the study.
5. Patients considered by the investigator to be able to complete themselves questionnaires used in the current study.
6. Signed Patient's Information Sheet and Informed Consent Form.

Patients with previously diagnosed COPD must meet all the following inclusion criteria:

1. Male and female of any age who were diagnosed with COPD before the study starts.
2. Patients whose COPD was not the direct reason for visiting the doctor or COPD patients who have COPD symptoms or signs requiring diagnostic or therapy.
3. Patients judged by the investigator as being capable to complete themselves the questionnaires used in the current study
4. Patient was scheduled to have the spirometry test performed in accordance with the existing medical practice before inviting him/her into the study
5. Signed Patient's Information Sheet and Informed Consent Form.

Exclusion criteria for patients with COPD risk factors:

1. Previously diagnosed chronic obstructive pulmonary disease.
2. Patients diagnosed with asthma, pulmonary tuberculosis, congenital lung abnormality, cystic fibrosis, lung cancer or cancer of the upper respiratory tract, patients who had a lung resection in the past due to pulmonary tuberculosis and other lung surgery, patients with stenosis of the upper respiratory tract, post-tracheotomy patients with the developed fibrotic stenosis of the trachea or post-intubation trachea stenosis, patients with ribs fractures of <3 weeks, pneumo- and hydrothorax of any etiology.
3. Patients who have contraindications for performing spirometry tests, patients with acute coronary syndrome or unstable circulatory dynamics. Patients who need emergency medical care at the moment of the visit.
4. Participation in any interventional clinical trial within 3 months prior the enrollment into the study and at the moment.

Patients with previously diagnosed COPD must meet all the following inclusion criteria:

1. Patients diagnosed with asthma, pulmonary tuberculosis, congenital lung abnormality, cystic fibrosis, lung cancer or cancer of the upper respiratory tract, patients who had a lung resection in the past due to pulmonary tuberculosis and other lung surgery, patients with stenosis of the upper respiratory tract, post-tracheotomy patients with fibrotic stenosis of the trachea or post-intubation trachea stenosis, patients with rib fractures of <3 weeks, pneumo- and hydrothorax of any etiology.
2. Active exacerbation of chronic obstructive pulmonary disease at the moment of enrollment into the study.
3. Patients who have contraindications for performing spirometry tests, patients with acute coronary syndrome or unstable hemodynamics. Patients who need emergency medical care at the time of the visit.
4. Participation in any interventional clinical trial within 3 months prior the enrollment into the study and at the moment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with COPD risk factors and patients with previously diagnosed COPD who have been observed in outpatient medical institutions of the RF are planned to be enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 4232 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The number of COPD cases first-time identified by the spirometry in relation to the total number of patients who visited the outpatient institutions of the RF during the study | Up to 5 months
Percentage of prescriptions for patients with COPD that correspond to the severity of the condition of the patients according to GOLD classification and GOLD recommendations for the treatment choice | Up to 5 months
Distribution (%) of patients with COPD who contacted the primary care doctors during the study based on bronchial obstruction severity (GOLD 1-4) and classes according to GOLD classification (2014) | Up to 5 months

SECONDARY OUTCOMES:
The percentage (%) of patients who contact the medical institutions of RF daily can be referred to the group with risk of COPD development | Up to 5 months
Score on SGRQ at 1st Visit in COPD patients receiving monotherapy with inhaled long-acting and super long-acting bronchodilators and in patients who are treated with combined drugs containing inhaled corticosteroids and long-acting β2 agonists | Up to 5 months
Score on САТ at 1st Visit in COPD patients receiving monotherapy with inhaled long-acting and super long-acting bronchodilators and in patients who are treated with combined drugs containing inhaled corticosteroids and long-acting β2 agonists | Up to 5 months
Mean number of puffs of SABA for 24h in COPD patients receiving monotherapy with inhaled long-acting and super long-acting bronchodilators and in patients treated with combined drugs (inhaled corticosteroids and long-acting β2 agonists) | Upto 5 months
The percentage of COPD patients in the routine practice of these medical institutions | Up to 5 months
Health-related economic losses calculated on the basis of the collected data (number of hospitalizations due to COPD exacerbations, calls of emergency service due to COPD, seeking outpatient care due to COPD) for the previous year | Up to 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Bedenkov, Study Director — AstraZeneca; Vladimir Archipov, Prof., Principal Investigator — I.M. Sechenov First Moscow State Medical University
Locations (22):
- Russia (22):
  - Research Site, Barnaul, Nis-rru-xxx-2014/2
  - Research Site, Blagoveshchensk, Nis-rru-xxx-2014/2
  - Research Site, Chelyabinsk, Nis-rru-xxx-2014/2
  - Research Site, Cherepovets, Nis-rru-xxx-2014/2
  - Research Site, Izhevsk, Nis-rru-xxx-2014/2
  - Research Site, Kazan', Nis-rru-xxx-2014/2
  - Research Site, Kemerovo, Nis-rru-xxx-2014/2
  - Research Site, Krasnoyarsk, Nis-rru-xxx-2014/2
  - Research Site, Moscow, Nis-rru-xxx-2014/2
  - Research Site, Naberezhnye Chelny, Nis-rru-xxx-2014/2
  - Research Site, Novosibirsk, Nis-rru-xxx-2014/2
  - Research Site, Omsk, Nis-rru-xxx-2014/2
  - Research Site, Petrozavodsk, Nis-rru-xxx-2014/2
  - Research Site, Ryazan, Nis-rru-xxx-2014/2
  - Research Site, Saint Petersburg, Nis-rru-xxx-2014/2
  - Research Site, Smolensk, Nis-rru-xxx-2014/2
  - Research Site, Tomsk, Nis-rru-xxx-2014/2
  - Research Site, Ulan-Ude, Nis-rru-xxx-2014/2
  - Research Site, Vladivostok, Nis-rru-xxx-2014/2
  - Research Site, Yakutsk, Nis-rru-xxx-2014/2
  - Research Site, Yfa, Nis-rru-xxx-2014/2
  - Research Site, Stavropol, Nis-rru-xxx-2014/3

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3275&filename=SUPPORT_REPORTSynopsis_2015-12-07.pdf